CLINICAL TRIAL: NCT00142636
Title: Coronary Artery Calcification in Chronic Kidney Disease Using Multidetector Row Spiral Computed Tomography
Brief Title: CRICKET Study, Coronary Calcium Scores in Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: PI/study contacts no longer at Institution
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Genzyme, a Sanofi Company (Industry)
Other Study IDs: CIP #S-03-133; CRADA CIP # S-03-133
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kideny Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Patients with Chronic Kidney Disease (CKD) have been shown to have high coronary calcium scores (CAC), but the temporal association between Glomerular Filtration Rate, CVD risk factors and CAC has not been described. This is a single-center, longitudinal, observational study. Subjects included adults aged 18 years to 65 years old without preexisting coronary artery disease (CAD). The CKD subjects (GFR < 60 ml/min) and the control subjects (GFR >/=60ml/min) were recruited. Laboratory measurements and MDCT scan were performed at baseline and after 12 months. Baseline CAC and average intact parathyroid hormone (iPTH) level were significantly greater in the CKD group. Baseline CAC scores of the CKD group were twice the value of the control group; however, CAC scores over one year were unchanged from baseline.

DETAILED DESCRIPTION:
Patients with Chronic Kidney Disease (CKD) have been shown to have high coronary calcium scores (CAC), but the temporal association between Glomerular Filtration Rate, CVD risk factors and CAC has not been described. This is a single-center, longitudinal, observational study. Subjects included adults aged 18 years to 65 years old without preexisting coronary artery disease (CAD). The CKD subjects (GFR < 60 ml/min) were recruited from the Nephrology Clinic, and the control subjects (GFR >/=60ml/min) were recruited from the Internal Medicine Clinic. Laboratory measurements and MDCT scan were performed at baseline and after 12 months. Baseline CAC and average intact parathyroid hormone (iPTH) level were significantly greater in the CKD group. Baseline CAC scores of the CKD group were twice the value of the control group; however, CAC scores over one year were unchanged from baseline. These observations suggest that CAC begins in earlier stages of CKD. Moreover, novel CVD risk factors including iPTH may accelerate CAD progression in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female ages 18 to 65 years
* Chronic Kidney disease patients, GFR <60mL/min as defined by MDRD (Levey) formula.
* Healthy volunteer controls, GFR >/= 60 mL/min
* Signed, written informed consent

Exclusion Criteria:

* Ages <18 or >65 years
* Pregnant subjects
* Subjects with history of severe obstructive pulmonary disease, CHF, stroke, arrythmia.
* Dialysis and kidney transplant patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-02; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Dylan E Wessman, M.D., Principal Investigator — Naval Medical Center, San Diego, Department of Internal Medicine
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Result] Dylan Wessman, M.D., Sandra Gilbert, Frank Mullens, M.D., Robin Parker, M.D., John Hammes, M.D., Lou Brenner, M.D. and Amit Sharma, M.D.